CLINICAL TRIAL: NCT05902559
Title: Assessment of Novel Biomarkers in Participants Undergoing Targeted Lung Health Checks
Acronym: ALPINE
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 155581
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low-dose CT (LDCT) screening for lung cancer (LCS) has been shown to reduce lung cancer specific mortality in multiple randomised controlled trials. However, although LDCT screening has been demonstrated to reduce cancer- specific mortality, there remain outstanding questions regarding how screening can be implemented. In particular, indeterminate nodules are common, and can be challenging to distinguish from benign nodules on CT appearances alone. Furthermore, distinguishing cancers which are likely to become clinically significant from those that will remain indolent is challenging, but essential to prevent over-treatment and overdiagnosis. There is significant interest in using a multi-modal approach to LCS, incorporating biomarkers obtained from minimally-invasive samples alongside LDCT to improve ability to recognise clinically-significant lung cancers at an early stage.

The Targeted Lung Health Check (TLHC) programme is an NHS programme with the aim of using LDCT screening in appropriately high-risk individuals to improve early diagnosis and survival in lung cancer. The North Central London TLHC programme started in December 2022.

The purpose of the ALPINE study is to develop a platform to allow collection of minimally-invasive samples from participants undergoing screening within the North Central London TLHC programme. The use of such biomarkers in the diagnosis of lung cancer is a rapidly developing field and novel techniques and technologies are continuously under development. The ALPINE study will generate a cohort with matched biosamples, CT scans and clinical data which will be uniquely well placed to serve to develop or validate biomarkers in lung cancer screening and risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Attended one of more visits as part of the NCL NHS TLHC programme
* Adults aged between 55 years and 74 years and 364 days
* Have capacity and can provide written consent

Exclusion Criteria:

* Declines participation in ALPINE
* Lacking capacity and unable to provide written consent
* Patients who are considered by the clinician to be unfit/not suitable for enrolment in ALPINE

Ages: 55 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants eligible for Low Dose CT scan screening in the North Central London Targeted Lung Health Check programme
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
To identify novel molecular, immune and clinical biomarkers to improve the sensitivity and specificity of lung cancer screening beyond what is achieved with conventional risk prediction models and low-dose CT scanning. | 5 years
  This includes proteomics, metabolomics, genomics and immune repertoire characterization performed on peripheral bloods.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No